CLINICAL TRIAL: NCT05537129
Title: A Prospective, Multicentral, Open-label, Randomized, Controlled Clinical Trial to Compare the Survival, Morbidity and Mortality of Laparoscopic and Open Total Gastrectomy for Gastric Cancer
Brief Title: Laparoscopic vs Open Total Gastrectomy for Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, PHD,MD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOTGGC
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer, Laparoscopic Total Gastrectomy, Open Total Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Total Gastrectomy (Experimental)
  Interventions: Procedure: Total Gastrectomy
- Open Total Gastrectomy (Active Comparator)
  Interventions: Procedure: Total Gastrectomy

INTERVENTIONS:
Procedure: Total Gastrectomy — The laparoscopic or open total gastrectomy with D2 lymphadenectomy was performed according to the Japanese gastric cancer treatment guidelines.

SUMMARY:
The aim of the present study is to demonstrated the the safety and feasibility of laparoscopic total gastrectomy comparing with open total gastrectomy.

DETAILED DESCRIPTION:
Gastric cancer is most common cause of cancer-related deaths in the world. Laparoscopic distal gastrectomy has been demonstrated to be safe and effective compared with open distal gastrectomy. With an increase in incidences of proximal gastric cancer over the last decades, total gastrectomy has been prefered by surgeons, and laparoscopic total gastrectomy has become the alternative option. However, the safety and feasibility of laparoscopic total gastrectomy have yet to be proved completely.

ELIGIBILITY:
Inclusion Criteria:

1. histologically proven gastric adenocarcinoma in the upper or middle third of the stomach (by preoperative gastrofiberscopy)
2. age between 20 and 80 years old
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. clinical stage I-III (T1-4aN0-2M0) according to the 8th edition of the Americal Joint Committee on Cancer System (Clinical stage was determined based on the finding of gastrofiberscopy and abdominal computed tomography)
5. scheduled for total gastrectomy with D2 lymphadenectomy, and possible for R0 surgery by this procedures (Lymphadenectomy is performed on the basis of the criteria of the Japanese
6. written informed consent
7. without preoperative chemotherapy and radiotherapy

Exclusion Criteria:

1. clinical stage T1-4N3M0 or T4bN0-3M0 according to the 8th edition of the Americal Joint Committee on Cancer System
2. history of chemotherapy, radiotherapy, immunotherapy or target therapy
3. perigastric lymphnode≥3cm
4. received gastric surgery (i.e. gastrectomy or gastrojejunostomy)
5. multiple primary tumors
6. suffering from other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, complicated by poorly controlled hypertension, diabetes, mental disorders or diseases.
7. patients need emergency operation with complication of gastric cancer
8. adhesion due to the previous intraabdominal surgery
9. need for combined organ resection due to aggression of gastric cancer of other disease,
10. vulnerable people who cannot communicate or are pregnant (or planning to be pregnant)
11. currently participating or participated in other clinical trials in the last 6 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
3 year-DFS | 3 year
  3 year-disease free survival

SECONDARY OUTCOMES:
3 year-OS | 3 year
  3 year-overall survival
morbidity and mortality rates | 30 days following surgeries
  morbidity and mortality within 30 days following surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Xu, PHD,MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No